CLINICAL TRIAL: NCT02471885
Title: A Single Centre Double-blinded Randomized Placebo Controlled Pilot Study Investigating the Effect of Remote Ischaemic preConditioning in ONCology Patients Undergoing Chemotherapy (ERIC-ONC)
Brief Title: Effect of Remote Ischaemic Conditioning in Oncology Patients
Acronym: ERIC-ONC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15/0276
Record Dates: First submitted 2015-05-05; First posted 2015-06-15 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Cardiotoxicity
Keywords: remote ischaemic conditioning; remote ischemic conditioning; cardio-oncology; anthracycline; troponin; chemotherapy; myocardial reperfusion injury
MeSH Terms: conditions — Cardiotoxicity; Myocardial Reperfusion Injury | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischaemic conditioning (Experimental): Remote ischaemic conditioning in the form of a blood pressure cuff on upper arm inflated upto 200 mm Hg (or systolic BP + 20 mm Hg if low platelets e.g. 50-150 x10^9/L, skip remote ischaemic conditioning (RIC) if platelets < 50 x 10^9/L) for 5 minutes, then deflated to 0 mm Hg for 5 minutes, for 4 cycles before beginning of chemotherapy infusion. The entire pre-conditioning phase will last 40 minutes.
  Interventions: Procedure: Remote Ischaemic Conditioning
- Control (Placebo Comparator): Blood pressure cuff on upper arm inflated to 10 mm Hg for 5 minutes, then deflated to 0 mm Hg for 5 minutes, for 4 cycles before beginning of chemotherapy infusion. The entire control comparator will last 40 minutes
  Interventions: Other: Placebo

INTERVENTIONS:
Procedure: Remote Ischaemic Conditioning — each cycle of Remote Ischaemic Conditioning (RIC) consists of inflating a blood pressure cuff on the upper limb (arm) upto 200mm Hg (systolic BP + 20 mm Hg for low platelets, e.g. 50-150 x 10^9/L; skip RIC if platelets < 50 x 10^9/L) for 5 minutes, then deflated to 0 mm Hg for 5 minutes.
  Other Names: Remote Ischaemic PreConditioning; Remote Ischemic Conditioning
  Arms: Remote ischaemic conditioning
Other: Placebo — Sham control blood pressure cuff placement at 10 mm Hg for 5 minutes, then deflated to 0 mm Hg for 5 minutes.
  Other Names: Sham
  Arms: Control

SUMMARY:
Cancer survival has improved steadily due to earlier detection and treatment. Despite the established efficacy of anthracycline chemotherapy, its damaging effects on the heart (cardiotoxicity) limits treatment and confers acute and long term adverse cardiovascular consequences. Protective strategies for the heart (cardioprotection) with iron binders (chelation), heart rate (beta blockade) and blood pressure (renin angiotensin inhibition) medications have demonstrated promise in adult cancer patients, but these treatments are typically prescribed only after significant changes in heart chamber size and pumping ability are detected by imaging investigations (myocardial dysfunction).

Furthermore, these conventional therapies are constrained by important side effects that affect bone marrow, blood pressure, and the kidneys.

Remote ischaemic conditioning (RIC) protects the heart by activating cell survival pathways through brief repeated inflations and deflations of a blood pressure cuff to limit blood flow temporarily (noninjurious ischaemia). These innate survival mechanisms prevent part of the cellular injury that occurs during the ischaemia reperfusion cascade during a heart attack (myocardial infarction). Ischaemia reperfusion injury also shares common biochemical pathways with anthracycline cardiotoxicity, and thus RIC may be a novel form of nonpharmacological cardioprotection that can be applied when undergoing anthracycline chemotherapy.

The investigators propose a pilot single centre randomised controlled trial to investigate the effect of RIC on reducing heart muscle damage (myocardial injury) in anthracycline-treated cancer patients. The investigators will assess subclinical myocardial injury using high-sensitivity blood tests (troponin T levels) and advanced imaging techniques, monitor heart rhythm disturbances (cardiac arrhythmia) and analyse metabolic changes in urine and blood during chemotherapy, at specified time points, and follow up to 5 years after completing chemotherapy treatment).

DETAILED DESCRIPTION:
This pilot study aims to demonstrate whether remote ischaemic preconditioning (RIC), delivered as a nonpharmacological treatment via repeated inflations and deflations of a limb blood pressure cuff, can reduce subclinical myocardial injury from anthracycline chemotherapy. Chemotherapy cardiotoxicity is the dose limiting constraint in anthracycline chemotherapy regimens, and conventional drug treatments to prevent and treat it are limited by important interactions with blood pressure, kidney function or bone marrow function. The lifetime cancer risk is between 1 in 2 and 1 in 3 in the general population. Cancer treatment and survival has improved steadily 50% of patients now survive their initial cancer diagnosis, but approximately 25 to 50% of survivors will have abnormal cardiac function over the next twenty years. Historically, anthracycline chemotherapy dosing has been stratified to limit the incidence of clinical heart failure to around 5%. More recent studies have reported at least one third of anthracycline chemotherapy patients demonstrate a significant rise in Troponin levels as a blood biomarker of subclinical myocardial injury as well as documented evidence of biomarker rise even after a single cycle of chemotherapy, and thus the absolute threshold for myocardial injury may be lower and thus more prevalent than these conservative figures.

In standard dosing regimens, chemotherapy may be delayed or suspended in cancer patients based on the simplified measure of ejection fraction (EF) as a measure of cardiac systolic function. Conventional heart failure treatments such as betablockers or ACE inhibitors are usually prescribed only after a significant fall in EF, even though myocardial injury occurs long before this imprecise measurement changes. RIC has been shown to reduce myocardial injury and improve outcomes in elective and emergency percutaneous coronary intervention (PCI) and elective coronary artery bypass graft surgery (CABG). The common biochemical pathways in ischaemia reperfusion and anthracycline-induced cardiac myocyte injury suggest that RIC may be an unexplored nonpharmacological treatment to reduce myocardial injury for cancer patients.

This pilot study aims to demonstrate the effectiveness of RIC as an elegant noninvasive, nonmedicinal treatment to reduce myocardial injury in cancer patients, and therefore poses no significant ethical issues. RIC is known to be a safe intervention with no known significant adverse effects. Some patients have reported mild discomfort during cuff inflation. A small number have experienced minor skin bruising at the cuff site which is transient. There are no known long term adverse effects of RIC,

Recruitment Patients will be identified by their usual oncology team, and referred to the cardiology team based solely on known inclusion and exclusion criteria, which will ensure this process is free from undue influence.

The benefits of the study include an increase in the scientific understanding of how RIC may lead to a reduction in myocardial injury, as well as longitudinal documentation of myocardial injury in the form of blood biomarkers, ECG changes, metabolic changes, and novel imaging markers in cancer patients undergoing a common form of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult or teenage young adult cancer patients with capacity
* Anthracycline-regimen chemotherapy (de novo or re-challenge)
* Able to tolerate peripheral blood pressure arm cuff inflation

Exclusion Criteria:

* Recent myocardial infarction in previous 4 weeks
* previous diagnosis of dilated, hypertrophic cardiomyopathy, amyloid or Anderson-Fabry Disease
* peripheral vascular disease
* Chronic Kidney Disease (estimated glomerular filtration rate (GFR) < 30 ml/min)
* Taking sulphonylureas
* lymph node dissection patients will need BP cuff on contra-lateral arm
* Skip remote ischaemic conditioning (RIC) cycle if very low platelets (e.g. platelets < 50 x 10^9/L, can have RIC when platelet counts recover, as per protocol).

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-12-16 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
hs-Troponin T (hs-TnT) levels | at baseline, at 3-24 hours after end of infusion of each chemotherapy cycle, then at initiation of chemotherapy infusion (cycles 2-6, occurring at intervals of 3-weeks), then at 1-, 3-, 6-, 12- months follow up
  Biomarker of myocardial injury using high-sensitivity Troponin-T for above time points as serial measurements.

SECONDARY OUTCOMES:
Major Adverse Clinical Cardiovascular Event (MACCE) | 1-, 3-, 6-, 12- months follow up
  Major Adverse Cardiovascular Event (myocardial infarction, clinical heart failure requiring admission, life-threatening arrhythmia atrioventricular (AV) block requiring pacemaker, cardiac or cancer death)
Echocardiographic global longitudinal strain (GLS) | at baseline, then at 3- and 12- months follow up
  Echocardiographic longitudinal function (GLS %)
Incidence of cardiac arrhythmia | at start of infusion of cycle 5 chemotherapy
  two weeks ambulatory electrocardiographic (ECG) monitoring for atrial fibrillation, supraventricular tachycardia, ventricular tachycardia, atrioventricular block
Biomarker N-terminal pro-brain natriuretic peptide (NT-proBNP) | at 3- months follow up
  for heart failure / raised left atrial pressure
Micro ribonucleic acid (RNA) and mitochondrial de-oxyribonucleic acid (DNA) analysis | at baseline and at 3-months follow up
  Comparison of changes in micro ribonucleic acid (miRNA) and mitochondrial deoxyribonucleic acid (mtDNA), markers of protein expression at baseline (before) and at 3-months' follow up after completing chemotherapy regimen

CONTACTS AND LOCATIONS:
Overall Officials: Derek M Yellon, PhD FACC FAHA, Principal Investigator — University College, London; Malcolm Walker, MD FRCP, Principal Investigator — University College London Hospitals; Alison Macklin, Study Director — University College London Hospitals
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Candilio L, Malik A, Ariti C, Barnard M, Di Salvo C, Lawrence D, Hayward M, Yap J, Roberts N, Sheikh A, Kolvekar S, Hausenloy DJ, Yellon DM. Effect of remote ischaemic preconditioning on clinical outcomes in patients undergoing cardiac bypass surgery: a randomised controlled clinical trial. Heart. 2015 Feb;101(3):185-92. doi: 10.1136/heartjnl-2014-306178. Epub 2014 Sep 24. PMID 25252696
- [Background] White SK, Frohlich GM, Sado DM, Maestrini V, Fontana M, Treibel TA, Tehrani S, Flett AS, Meier P, Ariti C, Davies JR, Moon JC, Yellon DM, Hausenloy DJ. Remote ischemic conditioning reduces myocardial infarct size and edema in patients with ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2015 Jan;8(1 Pt B):178-188. doi: 10.1016/j.jcin.2014.05.015. Epub 2014 Sep 17. PMID 25240548
- [Background] Sloth AD, Schmidt MR, Munk K, Kharbanda RK, Redington AN, Schmidt M, Pedersen L, Sorensen HT, Botker HE; CONDI Investigators. Improved long-term clinical outcomes in patients with ST-elevation myocardial infarction undergoing remote ischaemic conditioning as an adjunct to primary percutaneous coronary intervention. Eur Heart J. 2014 Jan;35(3):168-75. doi: 10.1093/eurheartj/eht369. Epub 2013 Sep 12. PMID 24031025
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Davies WR, Brown AJ, Watson W, McCormick LM, West NE, Dutka DP, Hoole SP. Remote ischemic preconditioning improves outcome at 6 years after elective percutaneous coronary intervention: the CRISP stent trial long-term follow-up. Circ Cardiovasc Interv. 2013 Jun;6(3):246-51. doi: 10.1161/CIRCINTERVENTIONS.112.000184. Epub 2013 May 21. PMID 23696599
- [Derived] Mallouppas M, Chung R, Ghosh AK, Macklin A, Yellon DM, Walker JM. Anthracyclines and Biomarkers of Myocardial Injury: The Effect of Remote Ischemic Conditioning. JACC CardioOncol. 2023 May 2;5(3):343-355. doi: 10.1016/j.jaccao.2023.03.008. eCollection 2023 Jun. PMID 37397080
- [Derived] Chung R, Maulik A, Hamarneh A, Hochhauser D, Hausenloy DJ, Walker JM, Yellon DM. Effect of Remote Ischaemic Conditioning in Oncology Patients Undergoing Chemotherapy: Rationale and Design of the ERIC-ONC Study--A Single-Center, Blinded, Randomized Controlled Trial. Clin Cardiol. 2016 Feb;39(2):72-82. doi: 10.1002/clc.22507. Epub 2016 Jan 25. PMID 26807534
- See also: Hatter Cardiovascular Institute, UCL — http://www.hatter-cardiovascular-institute.co.uk/